CLINICAL TRIAL: NCT01149317
Title: Acupuncture to Decrease Disparities in Outcomes of Pain Treatment
Brief Title: Acupuncture for Chronic Pain
Acronym: ADDOPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Diane Mckee, Associate Professor, Dept of Family and Social Medicine, Albert Einstein College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2007-306; R21AT004543 (NIH)
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Chronic Pain
Keywords: acupuncture; health services research; chronic pain; health disparities
MeSH Terms: conditions — Chronic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): Weekly acupuncture treatment for up to 14 weeks
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Weekly acupuncture treatment for up to 14 weeks to augment usual care

SUMMARY:
Chronic pain is a significant public health problem, associated with impairments of physical and psychological functioning. While a third or more of the general population may suffer from chronic pain, it is often under recognized and under treated in health care settings. Low income and minority samples experience disparities in the prevalence of chronic pain, in perceived access to effective pain treatment, and in consultations for pain. A great deal of literature suggests that acupuncture offers potential benefit in the management of chronic pain, but it is rarely available to low income patients. The Acupuncture to Decrease Disparities in Outcomes of Pain Treatment (ADDOPT) project will introduce and evaluate the addition of acupuncture to the management of chronic pain for ethnically diverse, low-income primary care patients. The project represents a collaboration between the New York City Research and Improvement Networking Group (NYC RING), a practice-based research network dedicated to decreasing health disparities through primary care research, the Continuum Center for Health and Healing,The Swedish Institute School of Acupuncture, and Pacific College of Oriental Medicine. Our intervention will involve addition of weekly acupuncture sessions at 3 urban primary care practices. During training sessions at each practice, primary care providers will become familiar with acupuncture and indications for referral. Patients will be eligible if they experience chronic pain due to neck pain, back pain, or osteoarthritis. Our process evaluation, guided by Glasgow's REAIM framework, will assess barriers to implementation and adoption of the intervention in busy urban practices and acceptability to patients and providers. The investigators will employ a quasiexperimental design to assess primary outcomes (pain and quality of life) and obtain preliminary estimates of secondary outcomes (health care utilization and costs) of the intervention at each health center. This design will permit comparison across sites to discern practice level differences in uptake and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain due to osteoarthritis, back pain or neck pain; English or Spanish speaking

Exclusion Criteria:

* Active substance abuse; cognitive impairment; coumadin therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2008-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 1 mo pre-acupuncture and 6 mo

SECONDARY OUTCOMES:
Pain Free Days | pre-acupuncture and 6 mo
Pain Impact Questionnaire | 1 mo pre-acupuncture and 6 mo
Quality of Life | 1 mo pre-acupuncture and 6 mo

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Diane McKee, MD, MS, Principal Investigator — Albert Einstein College of Medicine; Benjamin Kligler, MD, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States